CLINICAL TRIAL: NCT06895577
Title: Neoadjuvant Chemoradiotherapy Plus Sintilimab for MSS, Locally Advanced Rectal Cancer: A Single-Center, Open-Label, Single-Arm, Phase 2 Trial
Brief Title: Neoadjuvant Chemoradiotherapy Plus Sintilimab for MSS, Locally Advanced Rectal Cancer-
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to errors in the previously submitted modification, we request to withdraw it and will submit a corrected update shortly.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-37
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; PD-1; neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant SCRT followed by Sintilimab plus CAPOX (Experimental): neoadjuvant SCRT followed by Sintilimab plus CAPOX
  Interventions: Drug: neoadjuvant SCRT followed by Sintilimab plus CAPOX

INTERVENTIONS:
Drug: neoadjuvant SCRT followed by Sintilimab plus CAPOX — SCRT (a total of 25 Gy in 5 days) followed by sintilimab (3mg/kg intravenous drip on day 1; every 3-week cycle for two cycles) combined with CAPOX (oxaliplatin 130 mg/m2 intravenous infusion over 2 h on day 1, capecitabine 1000 mg/m2 orally twice daily from day 1-14, in every 3-week cycle for two cycles) 1 week later.

SUMMARY:
This research investigates the efficacy and safety of combining Sintilimab, a PD-1 inhibitor, with neoadjuvant chemoradiotherapy (NCRT) in patients with locally advanced microsatellite-stable (MSS) rectal cancer. Given the limitations of current treatment strategies in achieving optimal clinical outcomes, this prospective, single-center, phase II clinical trial aims to improve pathological complete response (pCR) rates and overall survival (OS). The primary endpoint is pCR, with secondary endpoints including disease-free survival (DFS) and the incidence of treatment-related adverse events. This study seeks to provide insights into a novel treatment paradigm for MSS locally advanced rectal cancer, potentially offering improved therapeutic options for this patient population.

DETAILED DESCRIPTION:
Locally advanced rectal cancer (LARC) presents a complex treatment challenge, often requiring a multimodal approach to achieve optimal cure rates and improve survival. Currently, the combination of short-course radiotherapy (SCRT) and neoadjuvant chemotherapy has become a critical treatment strategy for LARC patients. Compared to conventional long-course radiotherapy (LCRT), SCRT is associated with a shorter treatment duration, typically lasting only five days, which facilitates rapid tumor shrinkage and minimizes surgical delays. This expedited treatment approach not only reduces the risk of postponing surgery but also improves the management of patients by minimizing fatigue and treatment-related side effects associated with longer regimens.

Despite the promising outcomes associated with SCRT and neoadjuvant chemotherapy, a significant proportion of patients still do not achieve satisfactory clinical responses to standard treatment regimens.

In recent years, the emergence of immune checkpoint inhibitors has revolutionized cancer treatment. In particular, PD-1 inhibitors such as Sintilimab have demonstrated significant antitumor activity across various solid tumors, notably in microsatellite instability-high (MSI-H) cancers. However, the potential benefits of these agents in microsatellite-stable (MSS) rectal cancer remain insufficiently explored.

This study aims to investigate the effects of combining Sintilimab with neoadjuvant chemotherapy and SCRT in a single-center, phase II trial for MSS locally advanced rectal cancer. By evaluating treatment responses and survival outcomes, we hope to provide a novel therapeutic option that enhances clinical efficacy for patients with LARC.

ELIGIBILITY:
Inclusion Criteria:

With my consent and signed informed consent, willing and able to comply with the planned visits, research treatment, laboratory tests, and other test procedures.

Age 18-75. Patients with a pathologically or cytologically confirmed adenocarcinoma of the rectum, all other histological types excluded.

The distance between the lower margin of the rectal tumor lesion and the anal margin <12 cm.

The physical status score (ECOG) of the Eastern Cooperative Oncology Group was 0-1 (see Appendix 1).

T3-4/N+ was evaluated by pelvic enhanced MRI. Had not received systemic anti-tumor therapy for colon cancer, including cytotoxic drugs, immune checkpoint inhibitor therapy, molecular targeted therapy, endocrine therapy, etc.

Appropriate organ function based on the following laboratory test values obtained during the screening period: white blood cell count ≥3 × 10^9/L, neutrophil count ≥1.5 × 10^9/L, platelet count ≥75 × 10^9/L, serum total bilirubin ≤1.5 × upper limit of normal (UNL), AST (SGOT) or ALT (SGPT) ≤2.5 × UNL, serum creatinine ≤1.5 × UNL.

Female subjects of reproductive age must undergo a negative serum pregnancy test within 3 days prior to the start of the study drug and be willing to use a medically approved highly effective contraceptive method (such as an IUD, contraceptive pill, or condom) during the study period and within 3 months after the last study drug administration; male subjects whose partners are women of reproductive age should be surgically sterilized or agree to use effective contraception during the study period and for 3 months after the last study dosing.

Willing and able to comply with research procedures and visit plans.

Exclusion Criteria:

Whole-body CT, MRI, or PET-CT confirms distant metastases (M1). Patients with complete intestinal obstruction, active bleeding, or perforation requiring emergency surgery.

The presence of other active malignancies in the past or at the same time (except malignancies that have received curative treatment and have been free of disease for more than 5 years or cancers in situ that can be cured by adequate treatment).

Thrombotic or embolic events (e.g., cerebrovascular accident, including transient ischemic attack, pulmonary embolism, and deep vein thrombosis) occurred in the 12 months prior to study entry.

Myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac dysfunction, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure in the 12 months prior to enrollment.

Systemic antibiotic use ≥7 days within 4 weeks prior to enrollment, or unexplained fever >38.5°C during screening or prior to first dosing (fever due to tumor could be included).

Had received major operations such as laparotomy, thoracotomy, laparoscopic resection of organs, or severe trauma within 2 months before enrollment (the surgical incision should be completely healed before enrollment in this clinical trial).

Known presence of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related disease.

The presence of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia).

Untreated active hepatitis (hepatitis B defined as HBV-DNA ≥500 IU/ml; hepatitis C defined as HCV-RNA above the lower detection limit of analytical methods) or co-infection with hepatitis B and hepatitis C.

A known or suspected history of allergy to any of the relevant drugs used in the study.

Pregnant or lactating women. Women of reproductive age who do not use effective non-hormonal contraception (or refuse to use it) or men who are likely to have children.

The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participating in the study or interfere with the study results, as well as patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 1 month after the surgery
  Pathological complete response will be evaluated with American Joint Committee on Cancer (AJCC) Cancer Staging

SECONDARY OUTCOMES:
Margin-free (R0) resection rate | Immediately after the surgery
Tumor regression grade | 1 month after surgery
  Grading Standards TRG 0: Complete regression - No identifiable tumor cells remain. The tumor is entirely necrotic (dead).
  TRG 1: Minimal regression - There are few viable tumor cells left. The tumor has significantly decreased in volume but is not completely gone.
  TRG 2: Moderate regression - The tumor shows a mixed pattern. There are some necrotic areas, but viable tumor cells are still present.
  TRG 3: Poor regression - The tumor remains largely intact, with only a small reduction in size. A significant number of viable tumor cells are still observable.
Number of participants with surgical complications | 30 days after surgery
3-year event-free survival rate | 3-year event-free survival rate
Local recurrence | 3 years after the surgery
  Defined as an intrapelvic recurrence following a primary rectal cancer resection, with or without distal metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No